CLINICAL TRIAL: NCT00991159
Title: A Phase 1, Placebo-Controlled, Randomized Study To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Following Single, Escalating, Intravenous Doses Of RN316 (PF-04950615) In Healthy Adult Subjects
Brief Title: A Study To Access The Safety And Tolerability Of RN316 (PF-04950615) When Administered To Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: B1481001; RN316-101
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Endocrinology; Hypercholesterolemia; Hyperlipidemia; Lipid Metabolism Disorders RN316 PF-04950615
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- RN316 (Experimental)
  Interventions: Biological: RN316

INTERVENTIONS:
Biological: RN316 — Single, escalating doses of RN316 administered IV. Doses planned for testing = 0.3, 1.0, 3.0, 6.0, 12.0, and 18.0 mg/kg.

SUMMARY:
The study is designed to determine the safety and tolerability of RN316 when administered intravenously to healthy adult subjects. This is the first time RN316 has been given to humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory men and women (of non-childbearing potential) ages 18 -70 inclusive.
* Baseline total cholesterol ≥ 200 mg/dl, baseline LDL ≥ 130 mg/dl.
* BMI 18.5 to 35, and body weight ≤150 kg, inclusive.

Exclusion Criteria:

* Evidence of clinically significant disease that may increase the risk to the subject of study participation or interfere with interpretation of results.
* Secondary hyperlipidemia.
* Subjects who have taken lipid lowering compounds within the past 12 months prior to dosing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single, escalating, intravenous infusions of RN316 administered to healthy adult subjects | Entire duration of study

SECONDARY OUTCOMES:
pharmacokinetics of RN316 in plasma after administration of single, escalating, intravenous infusions of RN316 to healthy adult subjects | Entire duration of study
pharmacodynamic effect (lipid-lowering) of single, escalating, intravenous doses of RN316 administered to healthy adult subjects | Entire duration of study
single dose immunogenicity | Entire duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Miami Gardens, Florida

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] Udata C, Garzone PD, Gumbiner B, Joh T, Liang H, Liao KH, Williams JH, Meng X. A Mechanism-Based Pharmacokinetic/Pharmacodynamic Model for Bococizumab, a Humanized Monoclonal Antibody Against Proprotein Convertase Subtilisin/Kexin Type 9, and Its Application in Early Clinical Development. J Clin Pharmacol. 2017 Jul;57(7):855-864. doi: 10.1002/jcph.867. Epub 2017 Feb 9. PMID 28181260
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481001&StudyName=A%20Study%20To%20Access%20The%20Safety%20And%20Tolerability%20Of%20RN316%20%28PF-04950615%29%20When%20Administered%20To%20Healthy%20Adult%20Subjects